CLINICAL TRIAL: NCT04970446
Title: The MIRO II Study: Microbial Restoration in Inflammatory Bowel Diseases
Brief Title: Microbial Restoration in Inflammatory Bowel Diseases
Acronym: MIRO II
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St Vincent's Hospital Melbourne (Other)
Collaborators: The Queen Elizabeth Hospital (Other); BiomeBank Adelaide (Unknown); The University of Queensland (Other); Monash University (Other)
Responsible Party: Principal Investigator, Michael Kamm, The MIRO II Study: Microbial Restoration in Inflammatory Bowel Diseases, St Vincent's Hospital Melbourne
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: StvincentsmelbourneMIROII
Record Dates: First submitted 2021-07-18; First posted 2021-07-21 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-01

CONDITIONS: Fecal Microbiota Transplantation; Crohn Disease; Inflammatory Bowel Diseases; Microbiome
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Intervention Model Description: Prospective, two clinical center, parallel-arm, randomised, double-blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomisation tables will be computer generated by an independent statistician. The indistinguishable aspect of the FMT syringes (colour, packaging) will ensure the blindness of both patients and physicians in charge.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FMT arm (Active Comparator): Anaerobically prepared, freeze-thawed faecal microbiota transplantation
  Interventions: Drug: Antibiotics; Dietary Supplement: Dietician designed diet; Drug: FMT
- Placebo arm (Placebo Comparator): Placebo liquid formulation (normal saline, glycerol, food colorant)
  Interventions: Drug: Antibiotics; Dietary Supplement: Dietician designed diet; Other: Placebo

INTERVENTIONS:
Drug: Antibiotics — All patients will receive a one week course of antibiotic therapy.
Dietary Supplement: Dietician designed diet — All patients will be recommended dietary modification 3 weeks prior to, and during, the study.
Drug: FMT — Anaerobically prepared stool. Dosing will vary according to mode of administration.
  Arms: FMT arm
Other: Placebo — Placebo will contain food colourant, 0.9% normal saline and glycerol.
  Arms: Placebo arm

SUMMARY:
This is a prospective, two-centre, double-blind, parallel-arm, randomised, placebo-controlled trial evaluating the impact of FMT on patients with active Crohn's disease.

DETAILED DESCRIPTION:
The study will be conducted in two parts. The first part will involve all patients undergoing an optimisation phase, followed by randomisation into either intervention or placebo arms of the induction phase of the study. For patients achieving a pre-determined clinical response threshold at week 8 they will be re-randomised into the maintenance phase of the trial for a further 44 weeks.

FMT will be anaerobically prepared, freeze-thawed for administration.

ELIGIBILITY:
Inclusion Criteria:

Active Crohn's disease

* Confirmed endoscopic active inflammation (unless isolated small bowel disease that is inaccessible by endoscopy in which case sonographic inflammation is sufficient) within 6 months of study entry AND
* CDAI score of 220-450 AND
* One of the following:

  * CRP ≥5mg/L
  * faecal calprotectin ≥100μg/g
  * inflammation on imaging (either intestinal ultrasound or magnetic resonance imaging)
* Willing and able to attend the study sites for regular endoscopic procedures.

Exclusion Criteria:

Active perianal or fistulising disease; Pregnant or intending to become pregnant within 12 months; Enteropathy or colitis other than Crohn's disease; Symptomatic intestinal stricture likely to require surgical treatment; Presence of a stoma; Presence of an ileoanal pouch; Total white cell count less than 3.0 x 109/L; Albumin less than 20g/L; Immunodeficiency (beyond that caused by immune suppressants used for the treatment of IBD) e.g. HIV or Common variable immune deficiency; Anaphylaxis/severe allergy to food; Thiopurine, methotrexate, biologic agent or small molecule inhibitors or aminosalicylates whose dose has been modified within the past two months, 1 month and two weeks of study entry, respectively; Prebiotic, probiotic or antibiotic therapy, or over-the-counter supplements therapy in the two weeks prior to study entry; Rectal topical Crohn's disease therapy in the 2 weeks prior to study entry; Prednisolone dose >20mg or budesonide dose >6mg; Unwilling or unable to taper corticosteroids to zero within 8 weeks of initial FMT; Active gastrointestinal infection; Alcohol consumption of a dependent nature; Primary sclerosing cholangitis; Any condition that the treating gastroenterologist deems to pose a theoretical risk to the patient undertaking FMT; Any patient that the treating clinicians feel is incapable of participating in the safe use of FMT.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Clinical response | Week 8
  CDAI decrease of ≥100 or CDAI<150

SECONDARY OUTCOMES:
Clinical remission | Week 8 and week 52 or Week 16 and week 60 (for open FMT group)
  CDAI <150
Endoscopic response | Week 8 and 52 or Week 16 and 60
  SES-CD reduction by 25% and 50%
Endoscopic remission | Week 8 and week 52 Week 16 and 60
  SES-CD ≤2 or absence of ulcers
Histological Remission | Week 8 and 52 or Week 16 and 60
  The absence of ulcers; the absence of acute inflammation histologically; one of either Geboes Score or Robarts Histology Index
Radiological remission | Week 8 and 52 or Week 16 and 60
  IUS (BWT <3mm and/or Limberg 0 or 1) or MRI (Wall thickness <4mm and no or minimal wall enhancement)
Biochemical response | Week 8 and 52 or Week 16 and 60
  Normalisation of CRP and faecal calprotectin (<50ug/g, <100ug/g, <150ug/g, <200ug/g, <250ug/g
Time to outcomes | Duration of trial
  Time taken to achieve clinical response or remission during induction and maintenance phases
Maintenance of clinical remission | Weeks 52 or 60
  CDAI <150
Sustained clinical remission | Weeks 52 or 60
  CDAI <150
Steroid-free clinical remission | Weeks 52 or 60
  Steroid-free clinical remission
Safety outcomes | Duration of trial
  Adverse events
Scientific outcomes | Week 8 and 52 or Week 16 and 60
  Comparison of genetic, microbiological, metabolic and immunologic factors in the responders with the non-responders

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Kamm, MD, Principal Investigator — St Vincents Hospital
Locations (1):
- St Vincents Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP
Time Frame: When data becomes available
Access Criteria: TBC

REFERENCES:
- [Derived] Fehily SR, Wright EK, Basnayake C, Wilson-O'Brien AL, Stanley A, Marks EP, Russell EE, Hamilton AL, Bryant RV, Costello SP, Kamm MA. Faecal microbiota transplantation in Crohn's disease: an Australian randomised placebo-controlled trial protocol. BMJ Open. 2025 Apr 19;15(4):e094714. doi: 10.1136/bmjopen-2024-094714. PMID 40254304